CLINICAL TRIAL: NCT01711684
Title: An Open Label Study Employing the Topical Immunomodulator Diphenylcyclopropenone in a Stabilized Gel to Treat Cutaneous Metastases
Brief Title: Treatment of Cutaneous Metastases With Diphenylcyclopropenone (DPCP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Patricia Gilleaudeau, Co-Investigator, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JKR-0788
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Neoplasm Metastasis; Melanoma
Keywords: Neoplasm Metastasis; Melanoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma | interventions — diphenylcyclopropenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diphenylcyclopropenone (DPCP) (Experimental): Subjects will have DPCP in a topical gel formulation applied to their cutaneous metastatic lesions.
  Interventions: Drug: Diphenylcyclopropenone (DPCP)

INTERVENTIONS:
Drug: Diphenylcyclopropenone (DPCP) — Topical application of study drug
  Other Names: Diphencyprone; DCP

SUMMARY:
Melanoma is a life-threatening cancer which poses a significant health burden, especially when metastatic or spreading to areas other than the original tumor growth. Although various treatment options are currently available for melanoma, melanomas that have metastasized widely to the skin pose a significant clinical challenge as the available therapies have limited effect. This study proposes the use of a topically applied compound named diphenylcyclopropenone (DPCP) which has been shown to be effective in treating melanoma patients whose diseases have spread widely throughout the skin. DPCP works by having a patient's own immune system, which is usually used to fight infections, attack cancerous cells. This compound has commonly been used to treat other conditions such as warts and hair loss throughout the world for many years and is known to cause limited side effects. Altering a patient's own immune system through topical treatments has also been shown to benefit patients with other cancers that have metastasized to skin such as breast cancer. In this study, the investigators will use DPCP to treat cutaneous metastases of various cancers including melanoma. Our overall intention is to get a better understanding of effective immune responses in the skin that may mediate metastatic cancer regression or cure.

DETAILED DESCRIPTION:
This is an open label study to determine the efficacy and mechanism(s) of the proprietary DPCP gel composition as a topical immunotherapeutic agent for the treatment of cutaneous metastases. This study is investigator initiated, carried out only at Rockefeller University and the Sponsor holds the IND and is providing the test agent. The products to be evaluated are 0.4% DPCP, in a non-volatile gel vehicle, and 0.04% DPCP in the same gel vehicle applied to the target lesions biweekly for 14 weeks. It is our goal to apply the study drug to all cutaneous metastatic lesions, but at the Investigator's discretion, certain lesions will be avoided if they are in particularly difficult locations such as around the eyes or on the lips. The estimated duration of the study is 142 days with 112 days of treatment followed by subject examination on Day 142. If DPCP is shown to cause resolution of lesions by this visit, there will be the possibility of continuing DPCP use as long as study medication continues to be provided to The Rockefeller University.

ELIGIBILITY:
Inclusion Criteria:

* male or female at least 18 years of age, up to 99 years of age
* able to give verbal and written informed consent
* clinically diagnosed cancer with multiple cutaneous metastases that are able to be biopsied. The subject may or may not be on concomitant cancer treatments/have internal metastases.
* for women of childbearing potential (WOCBP) or in men whose partners may become pregnant, willingness to use an acceptable method of contraception to prevent pregnancy for the duration of the study (while receiving study medication and for one month following the last dose of study medication). Acceptable forms of contraception are listed in the informed consent form.
* must have a negative urine pregnancy test (for WOCBP)
* must be willing and able to have the therapy applied by the investigator, must be willing and able to self-apply the therapy, and must be willing and able to comply with study instructions and return for required clinic visits.
* clinically diagnosed melanoma with multiple cutaneous metastasis that are able to be biopsied. The subject will be on concurrent PD-1 checkpoint inhibitor therapy (standard nivolumab or pembrolizumab, not on another clinical trial) and may or may not have internal metastasis.

Exclusion Criteria:

* subjects taking any of the following systemic or topical therapies within 4 weeks of enrollment: corticosteroids, immunosuppressants, and/or any other medications that may affect the outcome of the study
* subjects who have active localized or systemic medical conditions that, in the opinion of the investigator, would preclude or make unsafe their participation in the study
* subjects with any underlying diseases or dermatological conditions of the affected areas that require the use of interfering topical or systemic therapy
* subjects who are nursing mothers, pregnant, or planning to become pregnant at anytime during the course of the study or within 30 days of study completion
* subjects who are unable to comply with study procedures, communicate effectively, cooperate with the investigator, or are unable to understand the study
* history, physical, social, or lab findings suggestive of any medical or psychological condition that would, in the opinion of the PI, make the candidate ineligible for the study
* HIV positive as determined by self-reported history and/or a HIV point-of-care test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

PRIMARY OUTCOMES:
clinically evident inflammatory response elicited by DPCP and the clinically evident efficacy of DPCP to treat cutaneous metastases | Day 142

SECONDARY OUTCOMES:
histological and gene expression profiling of biopsy specimens | Day 142

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States